CLINICAL TRIAL: NCT05887635
Title: A Pilot Human Investigation of the Safety, Tolerability and Effectiveness of the Aqua Medical Circumferential RF Vapor (RFV) Ablation System for Duodenal Mucosal Ablation for the Management of Type-2 Diabetes Mellitus (STEAM T-2DM Pilot)
Brief Title: Study of Duodenal Mucosal RF Vapor Ablation in Subjects With Type-2 Diabetes Mellitus
Acronym: STEAM T-2DM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aqua Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLD-1021-SA
Record Dates: First submitted 2023-05-22; First posted 2023-06-05 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: Diabetes Mellitus Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Study arm- RF Vapor Ablation arm (Experimental): This is a single arm study. All enrolled patients will be included in this arm
  Interventions: Device: RF Vapor Ablation

INTERVENTIONS:
Device: RF Vapor Ablation — RF Vapor ablation of the duodenum

SUMMARY:
The purpose of this clinical study is to test the hypothesis that RF vapor ablation of the duodenal mucosa will result in improvement in glycemic parameters, without complications (bleeding/ stricture / perforation).

The main aims of the study are :

1. Evaluate the safety of the device and procedure based on the reported adverse events that occur.
2. Evaluate the effectiveness of the device and procedure by comparing change in HbA1c from baseline to 168 days post procedure.
3. Evaluate device tolerability based on pain scores reported by patients. The subject population for this study are adults (18-65 years of age) with type-2 diabetes mellitus. Study participation is 6 months for each patient.

The study is comprised of 5 phases: Screening, Run-in, RF Vapor ablation procedure, and Post-vapor ablation follow-up (up to 168 days), Identification and long term follow up of responders

ELIGIBILITY:
Inclusion Criteria:

1. Men and non-pregnant women 18-65 years of age
2. Diagnosed with T2D for at least 3 years and less than or equal to 10 years
3. HbA1C of 7.5 - 10% (59-86 mmol/mol)
4. BMI ≥ 24 and ≤ 40 kg/m2
5. On a minimum of 1 stable oral anti-diabetic medications with no changes in medication in the previous 3 months prior to study entry Note: For subjects on sulfonylurea (SU) glucose-lowering drugs for diabetes, the only SUs permitted in the study will be glipizide or glimepiride, and their doses below half maximum labeled dosing will not be an exclusion for study entry. Subjects unwilling to reduce the dose of SU at the run-in period will be excluded.
6. Agrees to use an additional glucose-lowering treatment (e.g., liraglutide, other OAD with the exception of glyburide), if recommended by the study Investigator in case of persistent hyperglycemia.
7. Able to comply with study requirements and understand and sign the Informed Consent Form

Exclusion Criteria:

1. Diagnosis of Type-1 Diabetes
2. History of diabetic ketoacidosis or hyperosmolar nonketotic coma.
3. Probable insulin production failure, defined as fasting C Peptide serum <1 ng/mL (333pmol/l).
4. Previous use of any types of insulin for >1 month (at any time, except for treatment of gestational diabetes).
5. Current use of injectable medications for diabetes (insulin, GLP-1RA).
6. Current use of glyburide, a sulfonylurea (SU) glucose-lowering drug for diabetes.
7. History of severe hypoglycemia (more than 1 severe hypoglycemic event, as defined by need for third-party assistance, in the last year).
8. Known autoimmune disease, including but not limited to celiac disease, duodenal Crohn disease or pre-existing symptoms of systemic lupus erythematosus, scleroderma or other systemic autoimmune connective tissue disorder.
9. Previous GI surgery that could limit treatment of the duodenum such as Billroth 2, Roux-en-Y gastric bypass, or other similar procedures or conditions. (Prior laparoscopic sleeve gastrectomy (LSG) will not be an exclusion)
10. History of chronic or acute pancreatitis.
11. History of diabetic gastroparesis.
12. Known active hepatitis or active liver disease.
13. Acute gastrointestinal illness in the previous 7 days.
14. Known history of severe irritable bowel syndrome, radiation enteritis or other inflammatory bowel disease, such as Crohn's disease.
15. Known history of a structural or functional disorder of the esophagus that may impede passage of the device through the gastrointestinal tract or increase risk of esophageal damage during an endoscopic procedure, including moderate-severe (Grade C or D) esophagitis, dysphagia due to achalasia or stricture/stenosis, esophageal varices, esophageal perforation, or any other disorder of the esophagus.
16. Upper gastrointestinal conditions such as active ulcers, polyps, varices, strictures, congenital or acquired duodenal telangiectasia
17. Current use of anticoagulation therapy (such as warfarin) that cannot be discontinued for 7 days before and 14 days after the procedure.
18. Current use of P2Y12 inhibitors (clopidogrel, prasugrel, ticagrelor) that cannot be discontinued for 14 days before and 14 days after the procedure.
19. Unable to discontinue non-steroidal anti-inflammatory drugs (NSAIDs) during treatment through 4 weeks following the procedure. Use of acetaminophen and low dose aspirin is allowed.
20. Use of systemic glucocorticoids (excluding topical or ophthalmic application or inhaled forms) for more than 10 consecutive days within 12 weeks prior to the baseline visit.
21. Use of drugs known to affect GI motility (e.g. Metoclopramide)
22. Use of weight loss medications such as Sibutramine (e.g. Meridia), Orlistat (e.g. Xenical), Phentermine or over-the-counter weight loss medications (prescription medication)
23. Currently taking, or unable to stop taking dietary supplements or herbal agents, including vitamin C or multivitamins containing vitamin C at >500 mg per day, multivitamins containing biotin (vitamin B7), and supplements for hair, skin, and nail growth. Multivitamins not containing biotin are permitted.
24. Significant cardiovascular disease, including known history of valvular disease, or myocardial infarction, heart failure, transient ischemic attack, or stroke within 6 months prior to the Screening Visit.
25. Mean of 3 separate blood pressure measurements >180 mmHg (systolic) or >100 mmHg (diastolic).
26. Estimated glomerular filtration rate (eGFR) ≤ 60 ml/min/1.73m2 (estimated by MDRD).
27. Known immunocompromised status, including but not limited to individuals who have undergone organ transplantation, chemotherapy, or radiotherapy within the past 12 months, who have clinically significant leukopenia, who are positive for the human immunodeficiency virus (HIV) or whose immune status makes the participant a poor candidate for clinical trial participation in the opinion of the investigator.
28. Active illicit substance abuse or alcoholism (>2 drinks/day regularly)
29. Active malignancy within the last 5 years (excluding non-melanoma skin cancers)
30. Women breastfeeding
31. Participating in another ongoing clinical trial of an investigational drug or device.
32. Any other mental or physical condition which, in the opinion of the study investigator, makes the participant a poor candidate for clinical trial participation.
33. Critically ill or has a life expectancy <3 years
34. Use of heart pacemaker or other electronic device implants
35. General contraindications to deep or conscious sedation, general anesthesia, high risk as determined by anesthesiologist (e.g., ASA score 4 or higher), or contraindications to upper GI endoscopy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-09-02 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Safety endpoint | 1 month
  Number of subjects with reported device or procedure related SAEs or UADEs.
Efficacy endpoint | 6 months
  Change in HbA1c from baseline to 168 days post procedure
Tolerability Endpoint: | 14 days
  Descriptive statistics on Visual Analogue Scale(VAS) pain scores

SECONDARY OUTCOMES:
Change in HbA1c at 84 and 168 days post procedure | 168 days
  Change in HbA1c (from baseline) at 84 and 168 days post procedure will be analyzed
Change in HbA1c by visit over time | 168 days
  Change in HbA1c by visit over time, comparing with baseline
Change in FPG from baseline to 84 and 168 days post procedure | 168 days
  Change in FPG from baseline to 84 and 168 days post procedure
Change in FPG change by visit over time (168 days post procedure) | 168 days
  Change in FPG change by visit over time (168 days post procedure)
Proportion of ablation-treated subjects with an HbA1c improvement from baseline at 168 days | 168 days
  Proportion of ablation-treated subjects with an HbA1c improvement from baseline at 168 days
Changes in HOMA-IR by visit over time (168 days post procedure). | 168 days
  Changes in HOMA-IR by visit over time (168 days post procedure) from baseline
Change in UACR from baseline to 24 weeks post procedure | 24 weeks
  Change in UACR from baseline to 24 weeks post procedure
Change in ALT and AST from baseline to 24 weeks post procedure. | 24 weeks
  Change in ALT and AST from baseline to 24 weeks post procedure.

OTHER OUTCOMES:
Long term follow up endpoints among responders: Change in HbA1c over time | 2 years
  Change in HbA1c over time
Long term follow up endpoints among responders: Change in Fasting Plasma Glucose (FPG) over time | 2 years
  Change in FPG across each visit over time
Long term follow up endpoints among responders: Proportion of ablation-treated subjects with improvement from baseline | 2 years
  Proportion of ablation-treated subjects with an HbA1c improvement from baseline at 2 years.
Long term follow up endpoints among responders: Changes in HOMA-IR | 2 years
  Changes in HOMA-IR by visit over time
Long term follow up endpoints among responders: Change in Urine Albumin Creatinine Ratio (UACR) | 2 years
  Changes in UACR from baseline to 2 years post procedure
Long term follow up endpoints among responders: Change in ALT and AST | 2 years
  Change in ALT and AST from baseline to 2 years post procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Clinica Colonial, Santiago, Chile

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Norton BC, Papaefthymiou A, Telese A, Neiponice A, Hoebel PB, Vignolo P, Rodriguez Grunert LA, Haidry R. Radiofrequency vapor ablation for duodenal mucosal ablation in the treatment of type 2 diabetes: results from the first-in-human pilot study. IGIE. 2025 Mar 31;4(2):110-119. doi: 10.1016/j.igie.2025.03.008. eCollection 2025 Jun. PMID 41646468